CLINICAL TRIAL: NCT00673036
Title: French Registry of Acute Coronary Syndrome With or Without ST Elevation
Brief Title: French Registry of Acute Coronary Syndrome
Acronym: Fast-MI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 04-1244
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Coronary syndrome; Myocardial infarction; French registry
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adults (female and male) with a acute coronary syndrome
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 60 ml of whole blood

SUMMARY:
The Fast-MI registry was designed to evaluate the "real world" management of patients with acute myocardial infarction (MI), and to assess their in-hospital, medium and long-term outcomes

DETAILED DESCRIPTION:
Primary objectives : compare survival following the admission to a USIC according to the terms of care

ELIGIBILITY:
Inclusion Criteria:

* admission within the 48 hours after the occurence of acute myocardial infarction (AMI)
* written informed consent for the DNA and serum databank

Exclusion Criteria:

* AMI occured within the 48 hours after therapeutic intervention (bypass, coronary angioplasty or other chirurgical intervention)
* diagnostic of AMI not confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients in a Unit of Coronary Intensive Care (USIC) for a acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 3750 (Actual)
Dates: Start 2005-10; Primary Completion 2017-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
All causes mortality at each follow-up period | 6 months, each year

SECONDARY OUTCOMES:
Cardiovascular mortality | 6 month, each year
validation of guidelines across the country | 6 month, each year
Pharmacogenetic and cardiovascular genetic studies associated to clinical outcomes | 6 month each year
Serum databank for evaluation of biomarkers in MI | 6 month each year

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DANCHIN, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- French Society of Cardiology, Paris, France

REFERENCES:
- [Background] Hasdai D, Lev EI, Behar S, Boyko V, Danchin N, Vahanian A, Battler A. Acute coronary syndromes in patients with pre-existing moderate to severe valvular disease of the heart: lessons from the Euro-Heart Survey of acute coronary syndromes. Eur Heart J. 2003 Apr;24(7):623-9. doi: 10.1016/s0195-668x(02)00742-x. PMID 12657220
- [Background] Randomised trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet. 1994 Nov 19;344(8934):1383-9. PMID 7968073
- [Background] Sacks FM, Pfeffer MA, Moye LA, Rouleau JL, Rutherford JD, Cole TG, Brown L, Warnica JW, Arnold JM, Wun CC, Davis BR, Braunwald E. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial investigators. N Engl J Med. 1996 Oct 3;335(14):1001-9. doi: 10.1056/NEJM199610033351401. PMID 8801446
- [Background] Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. Lancet. 2002 Jul 6;360(9326):7-22. doi: 10.1016/S0140-6736(02)09327-3. PMID 12114036
- [Background] GUSTO investigators. An international randomized trial comparing four thrombolytic strategies for acute myocardial infarction. N Engl J Med. 1993 Sep 2;329(10):673-82. doi: 10.1056/NEJM199309023291001. PMID 8204123
- [Background] Andersen HR, Nielsen TT, Rasmussen K, Thuesen L, Kelbaek H, Thayssen P, Abildgaard U, Pedersen F, Madsen JK, Grande P, Villadsen AB, Krusell LR, Haghfelt T, Lomholt P, Husted SE, Vigholt E, Kjaergard HK, Mortensen LS; DANAMI-2 Investigators. A comparison of coronary angioplasty with fibrinolytic therapy in acute myocardial infarction. N Engl J Med. 2003 Aug 21;349(8):733-42. doi: 10.1056/NEJMoa025142. PMID 12930925
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] Gustafsson I, Torp-Pedersen C, Kober L, Gustafsson F, Hildebrandt P. Effect of the angiotensin-converting enzyme inhibitor trandolapril on mortality and morbidity in diabetic patients with left ventricular dysfunction after acute myocardial infarction. Trace Study Group. J Am Coll Cardiol. 1999 Jul;34(1):83-9. doi: 10.1016/s0735-1097(99)00146-1. PMID 10399995
- [Background] Torp-Pedersen C, Kober L. Effect of ACE inhibitor trandolapril on life expectancy of patients with reduced left-ventricular function after acute myocardial infarction. TRACE Study Group. Trandolapril Cardiac Evaluation. Lancet. 1999 Jul 3;354(9172):9-12. doi: 10.1016/s0140-6736(98)09374-x. PMID 10406358
- [Background] Pedersen OD, Bagger H, Kober L, Torp-Pedersen C. Trandolapril reduces the incidence of atrial fibrillation after acute myocardial infarction in patients with left ventricular dysfunction. Circulation. 1999 Jul 27;100(4):376-80. doi: 10.1161/01.cir.100.4.376. PMID 10421597
- [Background] Hall AS, Murray GD, Ball SG. Follow-up study of patients randomly allocated ramipril or placebo for heart failure after acute myocardial infarction: AIRE Extension (AIREX) Study. Acute Infarction Ramipril Efficacy. Lancet. 1997 May 24;349(9064):1493-7. doi: 10.1016/s0140-6736(97)04442-5. PMID 9167457
- [Background] Koren MJ, Hunninghake DB; ALLIANCE Investigators. Clinical outcomes in managed-care patients with coronary heart disease treated aggressively in lipid-lowering disease management clinics: the alliance study. J Am Coll Cardiol. 2004 Nov 2;44(9):1772-9. doi: 10.1016/j.jacc.2004.07.053. PMID 15519006
- [Background] Long-Term Intervention with Pravastatin in Ischaemic Disease (LIPID) Study Group. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. N Engl J Med. 1998 Nov 5;339(19):1349-57. doi: 10.1056/NEJM199811053391902. PMID 9841303
- [Background] Global Use of Strategies to Open Occluded Coronary Arteries in Acute Coronary Syndromes (GUSTO IIb) Angioplasty Substudy Investigators. A clinical trial comparing primary coronary angioplasty with tissue plasminogen activator for acute myocardial infarction. N Engl J Med. 1997 Jun 5;336(23):1621-8. doi: 10.1056/NEJM199706053362301. PMID 9173270
- [Background] Danchin N, Vaur L, Genes N, Etienne S, Angioi M, Ferrieres J, Cambou JP. Treatment of acute myocardial infarction by primary coronary angioplasty or intravenous thrombolysis in the "real world": one-year results from a nationwide French survey. Circulation. 1999 May 25;99(20):2639-44. doi: 10.1161/01.cir.99.20.2639. PMID 10338456
- [Background] Danchin N, Vaur L, Genes N, Renault M, Ferrieres J, Etienne S, Cambou JP. Management of acute myocardial infarction in intensive care units in 1995: a nationwide French survey of practice and early hospital results. J Am Coll Cardiol. 1997 Dec;30(7):1598-605. doi: 10.1016/s0735-1097(97)00371-9. PMID 9385882
- [Background] Vaur L, Danchin N, Genes N, Dubroca I, Etienne S, Ferrieres J, Cambou JP. Epidemiology of myocardial infarction in France: therapeutic and prognostic implications of heart failure during the acute phase. Am Heart J. 1999 Jan;137(1):49-58. doi: 10.1016/s0002-8703(99)70459-x. PMID 9878936
- [Background] Hanania G, Cambou JP, Gueret P, Vaur L, Blanchard D, Lablanche JM, Boutalbi Y, Humbert R, Clerson P, Genes N, Danchin N; USIC 2000 Investigators. Management and in-hospital outcome of patients with acute myocardial infarction admitted to intensive care units at the turn of the century: results from the French nationwide USIC 2000 registry. Heart. 2004 Dec;90(12):1404-10. doi: 10.1136/hrt.2003.025460. PMID 15547013
- [Background] Danchin N, Blanchard D, Steg PG, Sauval P, Hanania G, Goldstein P, Cambou JP, Gueret P, Vaur L, Boutalbi Y, Genes N, Lablanche JM; USIC 2000 Investigators. Impact of prehospital thrombolysis for acute myocardial infarction on 1-year outcome: results from the French Nationwide USIC 2000 Registry. Circulation. 2004 Oct 5;110(14):1909-15. doi: 10.1161/01.CIR.0000143144.82338.36. Epub 2004 Sep 27. PMID 15451803
- [Background] Ferrieres J, Cambou JP, Gueret P, Boutalbi Y, Lablanche JM, Hanania G, Genes N, Cantet C, Danchin N. Effect of early initiation of statins on survival in patients with acute myocardial infarction (the USIC 2000 Registry). Am J Cardiol. 2005 Feb 15;95(4):486-9. doi: 10.1016/j.amjcard.2004.10.016. PMID 15695134
- [Background] Heidenreich PA, Alloggiamento T, Melsop K, McDonald KM, Go AS, Hlatky MA. The prognostic value of troponin in patients with non-ST elevation acute coronary syndromes: a meta-analysis. J Am Coll Cardiol. 2001 Aug;38(2):478-85. doi: 10.1016/s0735-1097(01)01388-2. PMID 11499741
- [Background] Franklin K, Goldberg RJ, Spencer F, Klein W, Budaj A, Brieger D, Marre M, Steg PG, Gowda N, Gore JM; GRACE Investigators. Implications of diabetes in patients with acute coronary syndromes. The Global Registry of Acute Coronary Events. Arch Intern Med. 2004 Jul 12;164(13):1457-63. doi: 10.1001/archinte.164.13.1457. PMID 15249356
- [Background] Steg PG, Iung B, Feldman LJ, Cokkinos D, Deckers J, Fox KA, Keil U, Maggioni AP. Impact of availability and use of coronary interventions on the prescription of aspirin and lipid lowering treatment after acute coronary syndromes. Heart. 2002 Jul;88(1):20-4. doi: 10.1136/heart.88.1.20. PMID 12067934
- [Background] Amar J, Chamontin B, Ferrieres J, Danchin N, Grenier O, Cantet C, Cambou JP. Hypertension control at hospital discharge after acute coronary event: influence on cardiovascular prognosis--the PREVENIR study. Heart. 2002 Dec;88(6):587-91. doi: 10.1136/heart.88.6.587. PMID 12433885
- [Background] Danchin N, Grenier O, Ferrieres J, Cantet C, Cambou JP. Use of secondary preventive drugs in patients with acute coronary syndromes treated medically or with coronary angioplasty: results from the nationwide French PREVENIR survey. Heart. 2002 Aug;88(2):159-62. doi: 10.1136/heart.88.2.159. PMID 12117845
- [Background] Zeller M, Cottin Y, Brindisi MC, Dentan G, Laurent Y, Janin-Manificat L, L'Huillier I, Beer JC, Touzery C, Makki H, Verges B, Wolf JE; RICO survey working group. Impaired fasting glucose and cardiogenic shock in patients with acute myocardial infarction. Eur Heart J. 2004 Feb;25(4):308-12. doi: 10.1016/j.ehj.2003.12.014. PMID 14984919
- [Background] Chambless L, Keil U, Dobson A, Mahonen M, Kuulasmaa K, Rajakangas AM, Lowel H, Tunstall-Pedoe H. Population versus clinical view of case fatality from acute coronary heart disease: results from the WHO MONICA Project 1985-1990. Multinational MONItoring of Trends and Determinants in CArdiovascular Disease. Circulation. 1997 Dec 2;96(11):3849-59. doi: 10.1161/01.cir.96.11.3849. PMID 9403607
- [Background] Marques-Vidal P, Ferrieres J, Metzger MH, Cambou JP, Filipiak B, Lowel H, Keil U. Trends in coronary heart disease morbidity and mortality and acute coronary care and case fatality from 1985-1989 in southern Germany and south-western France. Eur Heart J. 1997 May;18(5):816-21. doi: 10.1093/oxfordjournals.eurheartj.a015347. PMID 9152652
- [Derived] Fayol A, Schiele F, Ferrieres J, Puymirat E, Bataille V, Tea V, Chamandi C, Albert F, Lemesle G, Cayla G, Weizman O, Simon T, Danchin N; FAST-MI Investigators. Association of Use and Dose of Lipid-Lowering Therapy Post Acute Myocardial Infarction With 5-Year Survival in Older Adults. Circ Cardiovasc Qual Outcomes. 2024 May;17(5):e010685. doi: 10.1161/CIRCOUTCOMES.123.010685. Epub 2024 Apr 29. PMID 38682335
- [Derived] Garcia R, Marijon E, Karam N, Narayanan K, Anselme F, Cesari O, Champ-Rigot L, Manenti V, Martins R, Puymirat E, Ferrieres J, Schiele F, Simon T, Danchin N. Ventricular fibrillation in acute myocardial infarction: 20-year trends in the FAST-MI study. Eur Heart J. 2022 Dec 14;43(47):4887-4896. doi: 10.1093/eurheartj/ehac579. PMID 36303402
- [Derived] Dillinger JG, Achkouty G, Albert F, Muller G, Labeque JN, Moisson L, Morelle JF, Cottin Y, Pezel T, Lim P, Aissaoui N, Schiele F, Ferrieres J, Angoulvant D, Henry P, Puymirat E, Simon T, Danchin N; FAST-MI investigators. Deleterious synergistic effects of acute heart failure and diabetes mellitus in patients with acute coronary syndrome: Data from the FAST-MI Registries. Arch Cardiovasc Dis. 2022 May;115(5):264-275. doi: 10.1016/j.acvd.2022.02.004. Epub 2022 Mar 4. PMID 35304066
- [Derived] Schiele F, Puymirat E, Ferrieres J, Simon T, Fox KAA, Eikelboom J, Danchin N; FAST-MI investigators. The FAST-MI 2005-2010-2015 registries in the light of the COMPASS trial: The COMPASS criteria applied to a post-MI population. Int J Cardiol. 2019 Mar 1;278:7-13. doi: 10.1016/j.ijcard.2018.11.138. Epub 2018 Dec 3. PMID 30538057
- [Derived] Danchin N, Puymirat E, Cayla G, Cottin Y, Coste P, Gilard M, Goldstein P, Braun F, Belle L, Montalescot G, Ferrieres J, Schiele F, Simon T; FAST-MI Investigators. One-Year Survival After ST-Segment-Elevation Myocardial Infarction in Relation With Prehospital Administration of Dual Antiplatelet Therapy. Circ Cardiovasc Interv. 2018 Sep;11(9):e007241. doi: 10.1161/CIRCINTERVENTIONS.118.007241. PMID 30354592
- [Derived] Puymirat E, Riant E, Aissaoui N, Soria A, Ducrocq G, Coste P, Cottin Y, Aupetit JF, Bonnefoy E, Blanchard D, Cattan S, Steg G, Schiele F, Ferrieres J, Juilliere Y, Simon T, Danchin N. beta blockers and mortality after myocardial infarction in patients without heart failure: multicentre prospective cohort study. BMJ. 2016 Sep 20;354:i4801. doi: 10.1136/bmj.i4801. PMID 27650822
- [Derived] Puymirat E, Schiele F, Zeller M, Jacquemin L, Leclercq F, Marcaggi X, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Do randomized clinical trial selection criteria reflect levels of risk as observed in a general population of acute myocardial infarction survivors? The PEGASUS trial in the light of the FAST-MI 2005 registry. Int J Cardiol. 2016 Nov 15;223:604-610. doi: 10.1016/j.ijcard.2016.08.191. Epub 2016 Aug 16. PMID 27561167
- [Derived] Feldman L, Steg PG, Amsallem M, Puymirat E, Sorbets E, Elbaz M, Ritz B, Hueber A, Cattan S, Piot C, Ferrieres J, Simon T, Danchin N; FAST-MI investigators. Editor's Choice-Medically managed patients with non-ST-elevation acute myocardial infarction have heterogeneous outcomes, based on performance of angiography and extent of coronary artery disease. Eur Heart J Acute Cardiovasc Care. 2017 Apr;6(3):262-271. doi: 10.1177/2048872615626354. Epub 2016 Jan 12. PMID 26758543
- [Derived] Pouche M, Ruidavets JB, Ferrieres J, Iliou MC, Douard H, Lorgis L, Carrie D, Brunel P, Simon T, Bataille V, Danchin N. Cardiac rehabilitation and 5-year mortality after acute coronary syndromes: The 2005 French FAST-MI study. Arch Cardiovasc Dis. 2016 Mar;109(3):178-87. doi: 10.1016/j.acvd.2015.09.009. Epub 2015 Dec 23. PMID 26711546
- [Derived] Puymirat E, Lamhaut L, Bonnet N, Aissaoui N, Henry P, Cayla G, Cattan S, Steg G, Mock L, Ducrocq G, Goldstein P, Schiele F, Bonnefoy-Cudraz E, Simon T, Danchin N. Correlates of pre-hospital morphine use in ST-elevation myocardial infarction patients and its association with in-hospital outcomes and long-term mortality: the FAST-MI (French Registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction) programme. Eur Heart J. 2016 Apr 1;37(13):1063-71. doi: 10.1093/eurheartj/ehv567. Epub 2015 Nov 17. PMID 26578201
- [Derived] Donataccio MP, Puymirat E, Parapid B, Steg PG, Eltchaninoff H, Weber S, Ferrari E, Vilarem D, Charpentier S, Manzo-Silberman S, Ferrieres J, Danchin N, Simon T. In-hospital outcomes and long-term mortality according to sex and management strategy in acute myocardial infarction. Insights from the French ST-elevation and non-ST-elevation Myocardial Infarction (FAST-MI) 2005 Registry. Int J Cardiol. 2015 Dec 15;201:265-70. doi: 10.1016/j.ijcard.2015.08.065. Epub 2015 Aug 8. PMID 26301654
- [Derived] Aissaoui N, Puymirat E, Simon T, Bonnefoy-Cudraz E, Angoulvant D, Schiele F, Benamer H, Quandalle P, Prunier F, Durand E, Berard L, Blanchard D, Danchin N. Long-term outcome in early survivors of cardiogenic shock at the acute stage of myocardial infarction: a landmark analysis from the French registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction (FAST-MI) Registry. Crit Care. 2014 Sep 19;18(5):516. doi: 10.1186/s13054-014-0516-y. PMID 25246084
- [Derived] Danchin N, Puymirat E, Steg PG, Goldstein P, Schiele F, Belle L, Cottin Y, Fajadet J, Khalife K, Coste P, Ferrieres J, Simon T; FAST-MI 2005 Investigators. Five-year survival in patients with ST-segment-elevation myocardial infarction according to modalities of reperfusion therapy: the French Registry on Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) 2005 Cohort. Circulation. 2014 Apr 22;129(16):1629-36. doi: 10.1161/CIRCULATIONAHA.113.005874. Epub 2014 Mar 21. PMID 24657993
- [Derived] Puymirat E, Taldir G, Aissaoui N, Lemesle G, Lorgis L, Cuisset T, Bourlard P, Maillier B, Ducrocq G, Ferrieres J, Simon T, Danchin N. Use of invasive strategy in non-ST-segment elevation myocardial infarction is a major determinant of improved long-term survival: FAST-MI (French Registry of Acute Coronary Syndrome). JACC Cardiovasc Interv. 2012 Sep;5(9):893-902. doi: 10.1016/j.jcin.2012.05.008. PMID 22995875
- [Derived] Simon T, Taleb S, Danchin N, Laurans L, Rousseau B, Cattan S, Montely JM, Dubourg O, Tedgui A, Kotti S, Mallat Z. Circulating levels of interleukin-17 and cardiovascular outcomes in patients with acute myocardial infarction. Eur Heart J. 2013 Feb;34(8):570-7. doi: 10.1093/eurheartj/ehs263. Epub 2012 Sep 6. PMID 22956509
- [Derived] Puymirat E, Aissaoui N, Silvain J, Bonello L, Cuisset T, Motreff P, Bataille V, Durand E, Cottin Y, Simon T, Danchin N; FAST-MI investigators. Comparison of bleeding complications and 3-year survival with low-molecular-weight heparin versus unfractionated heparin for acute myocardial infarction: the FAST-MI registry. Arch Cardiovasc Dis. 2012 Jun-Jul;105(6-7):347-54. doi: 10.1016/j.acvd.2012.04.002. Epub 2012 Jun 27. PMID 22800719
- [Derived] Juilliere Y, Cambou JP, Bataille V, Mulak G, Galinier M, Gibelin P, Benamer H, Bouvaist H, Meneveau N, Tabone X, Simon T, Danchin N; FAST-MI Investigators. Heart failure in acute myocardial infarction: a comparison between patients with or without heart failure criteria from the FAST-MI registry. Rev Esp Cardiol (Engl Ed). 2012 Apr;65(4):326-33. doi: 10.1016/j.recesp.2011.10.027. Epub 2012 Feb 20. PMID 22357361
- [Derived] Simon T, Steg PG, Gilard M, Blanchard D, Bonello L, Hanssen M, Lardoux H, Coste P, Lefevre T, Drouet E, Mulak G, Bataille V, Ferrieres J, Verstuyft C, Danchin N. Clinical events as a function of proton pump inhibitor use, clopidogrel use, and cytochrome P450 2C19 genotype in a large nationwide cohort of acute myocardial infarction: results from the French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) registry. Circulation. 2011 Feb 8;123(5):474-82. doi: 10.1161/CIRCULATIONAHA.110.965640. Epub 2011 Jan 24. PMID 21262992
- [Derived] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083